CLINICAL TRIAL: NCT05841966
Title: Surgeon-performed Intraoperative Transoral Ultrasound in Patients With Suspected Head and Neck Squamous Cell Carcinoma of Unknown Primary: a Prospective Diagnostic Accuracy Study
Brief Title: Surgeon-performed Intraoperative Transoral Ultrasound for Cancer of Unknown Primary
Acronym: OP-CUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Martin Garset-Zamani, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Unknown Primary Transoral US
Record Dates: First submitted 2023-02-16; First posted 2023-05-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cancer of Unknown Primary Site; Unknown Primary Cancer; Unknown Primary, Squamous Cell Carcinoma
MeSH Terms: conditions — Neoplasms, Unknown Primary; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Transoral Ultrasound (Experimental): Transoral ultrasound of the tonsils and tongue base under general anesthesia.
  Interventions: Diagnostic Test: Transoral Ultrasound

INTERVENTIONS:
Diagnostic Test: Transoral Ultrasound — The tonsils and tongue base will be scanned transorally using high-frequency intraoperative ultrasound transducers. Direct contact with the tonsils through the mouth is achieved during general anesthesia.

SUMMARY:
Adult patients suspected of Squamous Cell Carcinoma of Unknown Primary (SCCUP) will be prospectively enrolled at a tertiary head & neck cancer center at Copenhagen University Hospital - Rigshospitalet, Copenhagen, Denmark. All patients will undergo Magnetic Resonance Imaging (MRI) and Positron Emission Tomography-Computerized Tomography (PET-CT) prior to examination in general anesthesia. During general anesthesia, Intraoperative Transoral Ultrasound (ITUS) will be performed prior to panendoscopy. Detected tumors will be registered with specified oropharyngeal sub-locations. Blinded to ITUS, a consultant head & neck surgeon will perform panendoscopy. After examination, the surgeon is unblinded to ultrasound results. Final histopathology results from location-specified biopsies performed will be used as reference standard. The overall detection rate will be compared between ITUS, panendoscopy, PET-CT and MRI with sensitivity and specificity analysis. Oropharynx sub-location specific detection rate of ITUS vs. panendoscopy will be compared with logistic regression analysis.

DETAILED DESCRIPTION:
A prospective diagnostic study examining patients with suspected SCCUP will be performed at the Department of Otorhinolaryngology & Head & Neck Surgery, Copenhagen University Hospital - Rigshospitalet, Denmark. This specialized cancer center is responsible for the surgical work-up for approximately half of suspected SCCUP patients in the Danish population of 5.8 million.

Standard work-up of patients with suspected SCCUP in Denmark consists of same-day clinical examination combined with high resolution video endoscopy with NBI, surgeon-performed neck ultrasound and fine-needle aspiration cytology (FNAC) of suspected lymph nodes with same-day results. Cytology results can be further tested for Human Papillomavirus (HPV), and patients are booked for panendoscopic examination under general anesthesia with frozen section biopsy. Pre-operative cross-sectional imaging to locate the primary tumor includes MRI and 18-F Fluordeoxyglucose (FDG) PET-CT.

Intraoperative transoral ultrasound

During general anesthesia and prior to panendoscopy, ITUS will be performed while a consultant head & neck surgeon performing panendoscopy is blinded. A Fujifilm Arietta 850 or Arietta 65 (Fujifilm, Tokyo, Japan), BK5000 (BK Medical ApS, Herlev, Denmark), or Samsung RS85 (Samsung Medison, Seoul, South Korea) ultrasound machines will be used. Small-footprint, high-frequency transducers such as the Arietta L51K linear-array intraoperative robot transducer attached to a forceps, the BK5000 "flexible hockey-stick" 18XL5s, or the Samsung RS85 LA3-22AI "hockeystick" will be used. A Boyle-Davis gag or laryngoscope will be used to visualize the tonsils (Figure 1), while the transducer is placed onto each tonsil in transverse and sagittal planes. The tongue base will be scanned by pulling the tongue anteriorly by an assistant and placing the transducer directly onto the tongue base. Alternatively, the tongue can be retracted with a video-laryngoscope while revealing the tongue base. The tongue base will be scanned from side to side in the sagittal plane. The tongue can then be pulled to either the left or right side to angle the probe obliquely for transverse imaging. If a tumor is suspected, the tumor location is registered in the following categories, including indication of right or left side:

* Tonsil cranial.
* Tonsil caudal.
* Glossotonsillar sulcus.
* Anterolateral tongue base.
* Anteromedial tongue base.
* Posterolateral tongue base.
* Posteromedial tongue base.
* "Other" oropharynx sub-locations, including anterior & posterior pharyngeal arches, soft palate, uvula, posterior oropharynx wall, and vallecula.

B-mode video clips of both tonsils and the tongue base will be recorded. Power doppler for suspected tumors and the contralateral side will be performed. If a well-defined lesion is seen, the greatest tumor diameter and if possible, three-dimensional size is measured. The grade of tumor suspicion will be rated on a 5-point Likert scale ranging from 0 (very low) to 5 (very high).

Panendoscopy Following ITUS, the surgeon will perform standard panendoscopy of the pharynx including palpation of the oral cavity and oropharynx, and high-resolution video endoscopy with NBI. If the surgeon suspects a tumor, the location is registered with the same categories as above. Tumor suspicion will be rated on a 5-point Likert scale ranging from 0 (very low) to 5 (very high). The surgeon will categorize visual findings such as ulcers, exophytic tumors, asymmetric tissue, vulnerable/bleeding mucosa, suspect vasculature on NBI, or no suspect visual findings. The surgeon will categorize palpatory findings as soft or firm. The clinically visualized or palpated greatest tumor diameter will be estimated. The surgeon is then unblinded to ultrasound results. After unblinding from ultrasound, the investigators will register whether further directed biopsies from ultrasound suspected location are performed.

If the primary tumor is not located during panendoscopy, patients will tonsillectomied and the tonsils will be sliced in 2mm slices by head & neck pathologists in search of the primary tumor. If the primary tumor is still unknown and the neck metastasis is HPV+, then patients are offered Transoral Robotic Surgery (TORS) with diagnostic tongue base mucosectomy. These tongue base specimens will also be sliced in 2mm slices and examined by head & neck pathologists. If the primary tumor is located in final histopathology from either tonsillectomies or tongue base mucosectomy, the location of the tumors will be compared to the initially registered suspected ultrasound locations from panendoscopy.

Medical chart data The patient's age, sex, alcohol, smoking, largest cervical lymph node size, cervical lymph node side (right/left), date of panendoscopy, date of conclusive histopathology results, and date of treatment initiation will be obtained from medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Cytology-verified cervical lymph node metastasis from squamous cell carcinoma in neck levels I-IV with HPV+ cytology.
* Booked for panendoscopic examination under general anesthesia.
* Pre-operative MRI and PET-CT available.

Exclusion Criteria:

* Unable to provide written informed consent.
* Unable to complete full surgical work-up including palatine- and lingual tonsillectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Increased detection rate by adding ITUS to panendoscopy | Within 2-4 weeks after panendoscopy.
  The difference in proportion of patients with SCCUP where a primary tumor location is correctly detected by ITUS but not detected with panendoscopy alone.

SECONDARY OUTCOMES:
Ultrasonographic features of primary tonsil and tongue base tumors | 1 year
  The echogenicity, shape and doppler flow pattern relative to the normal and contralateral tonsil tissue will be compared in biopsy-verified primary tumors.
Comparison of detection rate of ITUS, panendoscopy, combined ITUS+panendoscopy, MRI and PET-CT for locating the primary tumor. | 1 year
  The percentage of primary tumors located is compared between all of the above tests.

OTHER OUTCOMES:
Average time in minutes used to perform transoral ultrasound | 1 year
  Average operative time, including setup with mouth gags, to perform transoral ultrasound in general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Todsen, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Århus University Hospital, Department of Otorhinolaryngology, Head & Neck Surgery, Aarhus
  - Rigshospitalet, Department of Otorhinolaryngology, Head & Neck Surgery & Audiology, Copenhagen

IPD SHARING:
Plan to Share IPD: No